CLINICAL TRIAL: NCT05834634
Title: Ultrasound Changes of the Vagus Nerve in Patients With Parkinsonism
Status: Recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nourelhoda Ahmed Ahmed Haridy, Doctor, Assiut University
Other Study IDs: Ultrasound of vagus nerve
Record Dates: First submitted 2023-04-18; First posted 2023-04-28 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Parkinsonism
Keywords: Vagus nerve; Parkinsonism; Nerve ultrasound
MeSH Terms: conditions — Parkinsonian Disorders | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Patients with parkinsonism
  Interventions: Device: Ultrasound
- Group 2: Healthy age and sex matched controls
  Interventions: Device: Ultrasound

INTERVENTIONS:
Device: Ultrasound — The patients and controls will be scanned at the Neurophysiology unit of the Department of Neurology, Neurology, psychiatry and Neurosurgery hospital, Assiut university hospital. The acquisition of ultrasound images was performed using a Philips HD11XE imaging system with an L12-8 linear array probe. Cross-sectional area (CSA) of the right and left Vagus nerves in each subject, perimeter, echogenicity, and fascicular structure will be assessed and measured by tracing the nerve just inside its hyperechoic rim. The nerve will be seen on ultrasound B-mode near the bifurcation of the carotid artery, dorsal to the internal and common carotid arteries, as a structure that is hypoechogenic in the centre and more hyperechogenic on the periphery (24, 25). Both the carotid artery and the internal jugular vein served as anatomical landmarks (25). Two separate CSA measurements, with the probe repositioned for each measurement, will be taken and they will be averaged.

SUMMARY:
In this study, the investigators will assess the Vagus nerve in two groups: Group 1 which include patients with parkinsonism and group 2 which included age and sex matched healthy control. The aim of the study is: detecting the difference between both groups and correlating the changes in the Vagus nerve cross sectional area with the motor and non motor manifestations of parkinsonism

DETAILED DESCRIPTION:
Parkinsonism is a syndrome characterized by the presence of six cardinal motor characteristics: resting tremor, rigidity, bradykinesia, loss of postural reflexes, flexed posture, and freezing. These combined symptoms identify clinically definite, probable, and possible parkinsonism (1). The most common form of parkinsonism is Parkinson's disease (PD) (1). Other forms of parkinsonism included atypical parkinsonism as progressive supranuclear palsy (PSP), multiple system atrophy (MSA), and corticobasal syndrome (CBS). The former types of parkinsonism are neurodegenerative disorders. Vascular parkinsonism (VP) is another form attributed to vascular etiology (2).

PD is the second-most common neurodegenerative disorder that affects 2-3% of the population ≥65 years of age. The main manifestation of PD is a clinical hypokinetic rigid syndrome. Also, numerous non-motor symptoms (NMS), including autonomic symptoms, such as orthostatic hypotension, constipation and urinary incontinence, have been suggested as preclinical symptoms (3). Other NMS include sleep alterations, dementia, depression, and pain that may severely compromise the quality of life (4).

The main neuropathologic hallmark is the formation of cytoplasmic inclusions called α-synuclein-enriched Lewy bodies and Lewy neurites. These aggregations are found throughout the brain, most pronounced in the substantia nigra compacta (5, 6). Also, these aggregations are present in the peripheral nervous system, more specifically in the Vagus nerve, which plays a vital role in autonomic control (7, 8). In addition, the Vagus nerve may play a crucial role in PD pathogenesis as it was hypothesized that α-synuclein aggregates form in the enteric nervous system and spread to the CNS via the autonomic nervous system (9).

Neuromuscular ultrasound is a non-invasive tool that can visualize nerves and roots with high resolution and accuracy (10). A recent systematic review reported that in PD, there is a degree of Vagus nerve atrophy that may be detected by ultrasound; therefore, it can be utilized as a marker for Vagus nerve lesions. However, correlation studies are lacking between the findings and clinical manifestations of parkinsonism (11).

Several studies were conducted to examine vagal neuron loss by ultrasonography, but they reported contradictory results. For example, some studies discovered considerable atrophy of the Vagus nerves in PD patients (12-15). However, other studies found no difference between PD patients and healthy controls (16-19). In addition, the link between Vagus nerve atrophy and other atypical parkinsonism, MSA, PSP, and CBS has not been extensively studied (20).

The present study aims to detect ultrasound changes in the Vagus nerve in patients with parkinsonism, compare the findings with healthy control, and correlate these changes with the motor and non-motor manifestations.

ELIGIBILITY:
A) Inclusion Criteria:

* All patients fulfill the criteria of case definition of parkinsonism.
* Gender: both sexes are included.
* Willingness to participate in the study and to be subjected to the disease-related examinations and assessments.
* Willing and able to provide informed consent.

B) Exclusion Criteria:

* Patients unable to give informed consent.
* History of chronic psychiatric or other central nervous system pathology and other neurodegenerative disorder(s).
* Patients with previous surgery in proximity of the Vagus nerve (for example carotid endarterectomy or implantation of Vagus nerve stimulator).
* Patients with known systemic diseases (such as diabetes mellitus, vascular disease, and peripheral neuropathy).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: * Patients diagnosed with Parkinsonism including Parkinsons disease diagnosed according to the criteria of the UK British Brain Bank (21) and successive revision (22) attending the neurology outpatient clinic, Department of Neurology and Psychiatry, Assiut University hospital.
  * Age and sex matched healthy control group, will be recruited from the outpatient
Sampling Method: Non-Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Comparing vagus nerve diameter between healthy controls and patients with parkinsonism | 1 day
  Detecting the ultrasound changes in Vagus nerve in patients with parkinsonism in comparison to age and sex matched healthy control.

SECONDARY OUTCOMES:
Correlation of the Vagus nerve ultrasound changes with the motor and non-motor manifestations of parkinsonism | 1 day
  Identifying the correlation of the Vagus nerve ultrasound changes with the motor and non-motor manifestations in patients with parkinsonism

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed AR Ahmed, Principal Investigator — Assiut University; Nourelhoda AA Haridy, Principal Investigator — Assiut University
Locations (1):
- Assiut University, Asyut, Egypt